CLINICAL TRIAL: NCT06632704
Title: Assessing the Colgate Assist Handle Toothbrush in Individuals With Impairment of Hand Movement.
Status: Completed | Type: Observational
Sponsor: Colgate Palmolive (Industry)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: CRO-2024-04-MTB-ASSIST HANDLE-
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2024-10

CONDITIONS: Movement Disorders and Physical Impairments
Keywords: hand movement impairment
MeSH Terms: conditions — Movement Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Adults aged 18-70 yrs, if applicable, primary caregiver: The study population will consist of 26 participants, aged 18-70 years old and of record at Penn Dental Medicine.
  Interventions: Device: Colgate Toothbrush assist

INTERVENTIONS:
Device: Colgate Toothbrush assist — toothbrush handle assignment to all subjects; subjects will have a choice between two brush heads

SUMMARY:
User experiences of Colgate Assist Handle toothbrush as indicated by questionnaire and interview

DETAILED DESCRIPTION:
Video recording of tooth brushing technique Picture of toothbrush bristles after study period

ELIGIBILITY:
Inclusion Criteria:

* Individuals with specific movement disorders and physical impairments, such as, but not limited to, Parkinson disease, Huntington disease, multiple sclerosis, arthritis, cerebral palsy, stroke, and/or tremors that affect their ability to perform daily tasks, such as brushing their teeth.

Exclusion Criteria:

* Individuals with severe oral health issues such as oral cancer, ulcers, or severe periodontal disease.
* Individuals who are unable to open their mouth enough that it would prevent using a brushing device.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 26 participants, aged 18-70 years old and of record at Penn Dental Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
user experience | 1 week, 2 weeks and 3 weeks
  User experiences of Colgate Assist Handle toothbrush as indicated by questionnaire and interview Video recording of tooth brushing technique Picture of toothbrush bristles

CONTACTS AND LOCATIONS:
Overall Officials: Eugene M Ko, DDS, Principal Investigator — Deputy Director, Center for Clinical and Translational Research Clinical Associate Professor, Department of Oral Medicine
Locations (1):
- University of Pennsylvania school of Dental Medicine, Philadelphia, Pennsylvania, United States